CLINICAL TRIAL: NCT03685227
Title: A Closer Look at Yoga Nidra: Sleep Lab Analyses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Collaborators: Oregon Health and Science University (Other); University of Manitoba (Other)
Responsible Party: Principal Investigator, Erica Sharpe, Research Investigator/BRIDG Program Fellow, National University of Natural Medicine
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ES62018
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Electroencephalography; Electrocardiography; Respiratory Rate; Surveys and Questionnaires
Keywords: Yoga Nidra; Electroencephalography; Electrocardiography; Respiratory rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participant will lie quietly for 90 minutes. They will be allowed to sleep.
- Yoga Nidra (Experimental): Participant will practice yoga nidra (using a recording) during the first 30 minutes of the 90 minute measurement period. Then they will be allowed to sleep.
  Interventions: Other: Yoga Nidra

INTERVENTIONS:
Other: Yoga Nidra — This is a mind/body technique. Specifically, it is a guided meditation, performed while lying down.
  Arms: Yoga Nidra

SUMMARY:
This study is being conducted in order to understand more about how the body responds to a mind/body practice called yoga nidra. Results from this study will be used to inform the design of future studies that investigate the effects of yoga nidra on sleep quality and insomnia.

Yoga nidra is a simple guided meditation technique that involves lying still on a mattress while listening to a voice. Participants will follow simple instructions that involve becoming aware of their body and breath, as well as various memories, emotions, and images. This practice is not religious in nature. The investigators do not believe it will conflict with any religious beliefs. The goal of this practice is to help get rid of mental, physical and emotional tensions.

DETAILED DESCRIPTION:
This clinical trial explores the physiological effects of yoga nidra and its connection to sleep. The investigators will measure patterns in brainwave activity, respiration and heart rate variability using EEG, and two wireless devices: the Spire® breath monitor and the Bodyguard® HRV monitor. This study will also address feasibility questions related to credibility and acceptability, using self-report surveys, drop-out rates, and participant feedback. Twenty-two participants will be recruited using digital and paper advertisements throughout Portland and the National University of Natural Medicine (NUNM). Interested individuals will contact the study coordinator, and then complete a screening call. During this telephone screening, the study coordinator will ask general questions and use standardized surveys to exclude participants based on inclusion/exclusion criteria. Prospective participants who pass the telephone screening will then be invited for two visits to the Helfgott Research Institute. Each visit will involve informed consent, followed by the completion of two eligibility surveys, and several intake questionnaires. The measurement periods will involve: 10 minutes of baseline data collection, 30 minutes of lying quietly or listening to a recording of yoga nidra, and then 1 hour of resting comfortably. Participants will be allowed to fall asleep during this time and will be left alone in the room with the lights out during the entire intervention (after the first 10 minutes of baseline data collection). When finished, participants will complete a few short questionnaires before their departure. The first visit will involve lying quietly as a baseline control. At the second visit, half of the population will be randomly selected to do yoga nidra and half will complete the baseline control measurements again.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia severity index (ISI) score 8-21 (subthreshold to moderately severe clinical insomnia)
* Can understand a recording in English

Exclusion Criteria:

* prescription sleeping medications
* regular mind/body practice within last 6 months
* diagnosed depression (or Patient Health Questionnaire (PHQ-2 into PHQ-9) score above 10)
* diagnosed sleep apnea (or STOP-BANG Sleep Apnea Questionnaire score of 3 or more)
* excessive alcohol use
* cannabis use
* smoking
* stimulant use
* shift work
* fibromyalgia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Change in EEG power (uV^2/Hz) of alpha brainwaves (defined by frequencies between 8-12 Hz) measured from the occipital region of the scalp. | 90 minutes
  Average change in alpha power (from visit 1 to visit 2) will be compared for intervention and control groups. Other frequency bands (delta, beta, and theta) will be measured as well. EEG measurements will be collected from the F3, C3, and O1 locations on the scalp.

SECONDARY OUTCOMES:
Change in time to sleep onset | 90 minutes
  Average change in time to sleep onset (SOL) from visit 1 to visit 2, will be compared for intervention and control groups. The EEG montage follows American Academy of Sleep Medicine (AASM) guidelines for sleep measurement, and includes sensors placed in the following locations: ChinZ, Chin1, E1, E2, F3, C3, and O1, with (contralateral) reference and ground electrodes clipped onto the right and left earlobes, respectively.
Change in heart rate variability (HRV) parameters | 90 minutes
  The average change (visit 1 to visit 2) in two HRV parameters (root mean square of successive differences between normal-to-normal intervals (RMSSD, ms); and high frequency power (HF, ms^2)) will be compared for intervention and control groups.
Change in respiration rate | 90 minutes
  Average change in respiratory rate (visit 1 to visit 2) will be compared for intervention and control groups.
Feasibility: Credibility of Intervention | Rating will occur immediately after their visit
  After the intervention, participants will rate perceived credibility of the intervention for its use in producing sleep.
Feasibility: Acceptability of Intervention | Seven months
  Acceptability will be determined using recruitment and dropout rates

CONTACTS AND LOCATIONS:
Overall Officials: Erica Sharpe, PhD, Principal Investigator — National University of Natural Medicine (NUNM)
Locations (1):
- National University of Natural Medicine, Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sharpe E, Butler MP, Clark-Stone J, Soltanzadeh R, Jindal R, Hanes D, Bradley R. A closer look at yoga nidra- early randomized sleep lab investigations. J Psychosom Res. 2023 Mar;166:111169. doi: 10.1016/j.jpsychores.2023.111169. Epub 2023 Jan 29. PMID 36731199

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT03685227/Prot_SAP_000.pdf